CLINICAL TRIAL: NCT05869604
Title: Improving Cardiovascular Disease Risk Factors in Survivors of Adolescent and Young Adult Cancer With Obesity: Adaptation and Pilot Testing of a Behavioral Weight and Symptom Management Intervention
Brief Title: Healthy Lifestyles After Cancer for Adolescents and Young Adults: A Program to Reduce Cardiovascular Risk Factors
Acronym: HEALTHY-AYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00110049
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Cardiovascular Diseases; Weight Management; Pain; Fatigue; Distress, Emotional; Physical Inactivity
Keywords: AYA Cancer Survivors; Symptom management; Health Behavior Change
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Pain; Fatigue; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEALTHY AYA (Experimental): Participants randomized to the intervention arm will receive an 8 session intervention providing instruction in cognitive and behavioral symptom coping strategies as well as behavioral strategies to improve diet and decrease sedentary time.
  Interventions: Behavioral: HEALTHY AYA
- Education Control (Other): Participants randomized to the education control arm will receive information about topics of relevance to adolescent and young adult cancer survivors including sleep, cognitive problems, finances, sexual health, and return to work/school.
  Interventions: Other: Education Control

INTERVENTIONS:
Behavioral: HEALTHY AYA — 8-session health lifestyle behavior intervention combining behavioral symptom management strategies with strategies to improve diet and increase physical activity.
  Arms: HEALTHY AYA
Other: Education Control — Participants will receive paper materials on topics of relevance to adolescent and young adult cancer survivors.
  Arms: Education Control

SUMMARY:
There are close to 700,000 survivors of adolescent and young adult (AYA) cancer (aged 15 to 39 at diagnosis) in the US. Survivorship for AYAs is often complicated by long-term and late-effects. Cardiovascular disease (CVD), in particular, is a leading cause of death for cancer survivors and is a growing public health concern for survivors diagnosed as AYAs. Risk of CVD may be associated with treatment exposures and may be potentiated by weight gain and poor health behaviors. Healthy eating and physical activity are key behaviors for weight loss and maintenance and may be protective against CVD risk, yet few AYA cancer survivors adhere to guidelines for healthy eating or activity. AYA survivors' abilities to engage in health behaviors (i.e., healthy eating, physical activity) necessary to manage weight may also be challenged by persistent cancer-related symptoms (i.e., pain, fatigue, psychological distress). Thus, weight gain is common. Using input from AYA cancer survivors, the investigators have adapted a behavioral weight and symptom management protocol for AYA cancer survivors with obesity to create an intervention that is responsive to AYAs' unique needs. A pilot randomized controlled trial will be conducted to examine intervention feasibility and acceptability and to examine patterns of change in outcomes including weight, body mass index, symptoms (e.g., pain, fatigue, distress) as well as other CVD risk factors, including blood pressure, cholesterol (total, HDL, LDL), HbA1c, and atherosclerotic cardiovascular disease (ASCVD) risk score.

DETAILED DESCRIPTION:
There are close to 700,000 survivors of adolescent and young adult (AYA) cancer (aged 15 to 39 at diagnosis) in the US. Advances in treatment have yielded five year survival rates of >80% suggesting that the majority of AYAs will become long-term cancer survivors. While trends in survival are encouraging, the survivorship trajectories for AYAs are complicated by long-term and late-effects. Cardiovascular disease (CVD), in particular, is a leading cause of death for cancer survivors and is a growing public health concern for survivors diagnosed as AYAs. AYA cancer survivors have more than a two-fold risk of CVD when compared to age-matched peers and are at significantly greater risk of cardiac mortality. Risk of CVD may be associated with treatment exposures and may be potentiated by weight gain and poor health behaviors. Healthy eating and physical activity are key behaviors for weight loss and maintenance and may be protective against CVD risk. Adolescence and young adulthood are important developmental periods for the establishment of lifelong healthy behaviors, yet few AYA cancer survivors adhere to recommended guidelines for healthy eating or activity. Moreover, they report struggling to identify and maintain strategies to manage diet, improve nutrition, and increase activity. AYA survivors' efforts to engage in positive health behaviors (i.e., adhere to exercise and nutrition recommendations) necessary to manage weight may also be challenged by persistent cancer-related symptoms (i.e., pain, fatigue, psychological distress). Thus, weight gain is common, with >50% of AYA survivors classified as overweight or obese. Interventions for AYAs with obesity that aim to lower CVD risk through weight management, however, are rare and do not address symptoms that challenge healthy eating and activity despite recognition of the importance of improving health behaviors and symptom management in AYAs' transition to survivorship. The PI recently developed and evaluated a 12-session, in-person behavioral weight and symptom management intervention for breast cancer survivors with obesity and their intimate partners. Based on input from AYA cancer survivors, this intervention was adapted for AYA cancer survivors with obesity to produce an intervention responsive to AYAs' unique needs. A pilot RCT will be conducted to examine intervention feasibility and acceptability as well as patterns of change in outcomes. N=36 AYAs will be randomized to the intervention or education control arms. The protocol will be delivered via videoconferencing over 8 sessions. Assessments will be completed at baseline and post-treatment. AYAs will be weighed, have their blood pressure taken, complete a blood draw, and respond to self-report measures (e.g., symptoms, symptom interference, diet, activity). Weight and body mass index (BMI) will be assessed. Other CVD risk factors to be assessed include blood pressure, cholesterol (total, HDL, LDL), HbA1c, and atherosclerotic cardiovascular disease (ASCVD) risk score.

ELIGIBILITY:
Inclusion Criteria:

* History of cancer
* Diagnosed with cancer between the ages of 18 and 39
* Within 5 years of completing cancer treatments
* BMI >30
* Healthy enough to participate in home-based physical activity
* Able to speak and read English
* Able to provide informed consent

Exclusion Criteria:

* Current pregnancy
* Non-ambulatory
* Major mental illness (i.e., schizophrenia)
* untreated /uncontrolled mental illness (i.e., bipolar disorder)
* residence >60 miles from the research site

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of study recruitment | 12 months
  Number of participants recruited over the course of 12 months.
Session attendance | Following completion of the intervention (up to 3 months)
  Treatment feasibility will be assessed by measuring the session attendance rate for each participant.
Participant attrition | Following completion of the intervention (up to 3 months)
  Participant attrition will be assessed by measuring the number of participants who drop out of the study
Intervention acceptability: Treatment Acceptability Questionnaire | Following completion of the intervention (up to 3 months)
  The Treatment Acceptability Questionnaire is a six-item scale assessing participants' views of an intervention as acceptable, ethical, and effective.
  Items are rated on a 7-point Likert scale (e.g., 1 "very unacceptable" to 7 "very acceptable").
Intervention satisfaction: SSTS-R | Following completion of the intervention (up to 3 months)
  Intervention satisfaction will be assessed using the SSTS-R, a 13-item measure with the first 12-items on a five-point scale ranging from 1 "strongly disagree" to 5 "strongly disagree." The 13th item asks, "How much did the program help with the specific concern that led you to participate?" with 5 answer choices ranging from "made things a lot better" to made things a lot worse."
Open-Ended Questions About the Program | Following completion of the intervention (up to 3 months)
  Intervention will be evaluated using 3 open-ended questions, including the following: "1) What was the most helpful part of the program?," "2) What was the least helpful part of the program?", and "3) What suggestions do you have for us to help improve the program?"

SECONDARY OUTCOMES:
Change in diet and eating behavior: Three factor eating questionnaire | Baseline, follow-up assessment (up to 3 months)
  Eating behaviors will be assessed using the Three Factor Eating Questionnaire (TFEQ). The 21-item short-form will be used for the present study. The TFEQ measures three domains of eating behavior: 1) cognitive restraint, 2) uncontrolled eating, and 3) emotional eating.
Change in weight | Baseline, follow-up assessment (up to 3 months)
  Participants will be weighed at each assessment.
Change in diet: Dietary screener questionnaire | Baseline, follow-up assessment (up to 3 months)
  The Dietary Screener Questionnaire is a 25-item measure asking participants to rate on the frequency of eating/drinking certain foods in the last week.
Change in Physical Activity: Stanford L-Cat | Baseline, follow-up assessment (up to 3 months)
  The L-Cat is a measure of physical activity. Individuals identify which descriptive category best describes their level of activity during leisure time in the last month. Descriptive categories range from inactive to very active.
Change in Pain: Brief Pain Inventory (BPI) | Baseline, follow-up assessment (up to 3 months)
  The BPI is a 9-item self-report measure assessing pain severity. Participants rate their pain on a scale from 0 to 10 where 0 represents "no pain" and 10 represents "pain as bad as you can imagine." Participants also rate their level of interference from pain.
Change in Fatigue: PROMIS Fatigue Scale | Baseline, follow-up assessment (up to 3 months)
  The Promis Fatigue Scale is a 8-item self-report measure of fatigue in the last week. Participants are asked to respond to items (e.g., "I felt fatigued", "I have troubled starting things because I am tired") using scales ranging from 1 to 5.
Change in Depressive Symptoms: PROMIS Depression Short Form | Baseline, follow-up assessment (up to 3 months)
  Depressive Symptoms will be assessed using the PROMIS Depression Short Form, an 8-item measure assessing symptoms of depression in the last week. Participants are asked to respond to items (e.g., "I felt sad," "I felt helpless") using a five-point scale ranging from 1 "never" to 5 "always."
Change in Anxiety: PROMIS Anxiety Short Form | Baseline, follow-up assessment (up to 3 months)
  Symptoms of Anxiety will be assessed using the PROMIS Anxiety Short Form, an 8-item measure assessing symptoms of anxiety in the last week. Participants are asked to respond to items (e.g., "I felt nervous," "I felt tense") using a five-point scale ranging from 1 "never" to 5 "always".

OTHER OUTCOMES:
Change in Self-Efficacy: The Self-Efficacy for Managing Chronic Disease Scale | Baseline, follow-up assessment (up to 3 months)
  The Self-Efficacy for Managing Chronic Disease Scale is a 6-item scale. Participants rate their confidence in keeping pain, fatigue, emotional distress, and other symptoms from interfering with things they want to do on a scale from 1 "not at all confident" to 10 "totally confident."
Change in Self-Efficacy for weight management: Weight efficacy Lifestyle questionnaire- short form | Baseline, follow-up assessment (up to 3 months)
  The Weight Efficacy Lifestyle Questionnaire is an 8-item measure of eating self-efficacy. Participants are asked to provide information about how certain they are that they can resist overeating in difficult situation (e.g., over the weekend, when tired, etc.). Response choices range from 0= "not at all confident" to 10= "very confident."
Change in blood pressure (systolic and dyastolic) | Baseline, follow-up assessment (up to 3 months)
  Both systolic and dyastolic blood pressure will be assessed at the baseline and follow-up assessment.
Change in total cholesterol | Baseline, follow-up assessment (up to 3 months)
  Cholesterol will be assessed through peripheral blood at the baseline and follow-up assessment.
Change in LDL | Baseline, follow-up assessment (up to 3 months)
  LDL will be assessed through peripheral blood at the baseline and follow-up assessment
Change in HDL | Baseline, follow-up assessment (up to 3 months)
  HDL will be assessed through peripheral blood at the baseline and follow-up assessments.
Change in Triglycerides | Baseline, follow-up assessment (up to 3 months)
  Triglycerides will be assessed through peripheral blood at the baseline and follow-up assessments.
Concentration of HbA1c | Baseline, follow-up assessment (up to 3 months)
  HbA1c will be assessed through peripheral blood at the baseline and follow-up assessments.
Change in Atherosclerotic Cardiovascular Disease (ASCVD) risk | Baseline, follow-up assessment (up to 3 months)
  The 10 year risk for ASCVD is calculated using a patient's age, sex, race, systolic blood pressure, diastolic blood pressure, total cholesterol, HDL, LDL, history of diabetes, smoking status, whether or not they're on hypertension treatment, and whether or not they're on statin.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline S Dorfman, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No